CLINICAL TRIAL: NCT04449185
Title: Change of Gut Microbiome and Symptom After H.Pylori Eradication Therapy in Patients With Functional Dyspepsia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Kee Wook Jung, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0621
Record Dates: First submitted 2020-06-22; First posted 2020-06-26 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Dyspepsia
Keywords: Dyspepsia; Microbiome; Eradication therapy
MeSH Terms: conditions — Dyspepsia | interventions — tegoprazan; BID protein, human; Amoxicillin; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HP eradication group (Experimental): HP eradication group
  Tegoprazan 50mg bid + amoxicillin 1000mg bid + clarithromycin 500mg bid for 10 days
  Interventions: Drug: Tegoprazan 50mg bid + amoxicillin 1000mg bid + clarithromycin 500mg bid for 10 days

INTERVENTIONS:
Drug: Tegoprazan 50mg bid + amoxicillin 1000mg bid + clarithromycin 500mg bid for 10 days — Tegoprazan 50mg bid + amoxicillin 1000mg bid + clarithromycin 500mg bid for 10 days

SUMMARY:
The aims of the investigators' study are to investigate the effect of H.pylori eradication on the human gut microbiome and symptoms of functional dyspepsia.

DETAILED DESCRIPTION:
Accumulating evidence shows that Helicobacter pylori protects against some metabolic and immunological diseases in which the development of these diseases coincide with temporal or permanent dysbiosis. Helicobacter pylori eradication therapy has the potential to improve symptoms of functional dyspepsia. The aims of our study are to investigate the effect of H.pylori eradication on the human gut microbiome and symptoms of functional dyspepsia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who has diagnosed with functional dyspesia by Rome IV criteria

Exclusion Criteria:

* Known GI malignancy
* Previous Helicobater pylori eradication history
* Severe systemic disease
* Previous GI surgery
* Uncorrectable coagulopathy: INR > 1.5 or platelet < 50,000/ml
* Pregnant or breastfeeding women
* Atrophic gastritis, open type

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-06-30 (Estimated); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
Change of gut microbiome | at 3 months, and 6 months
  Change of gut microbiome at 3 months, and 6 months regardless of Helicobater positive or negative

SECONDARY OUTCOMES:
Symptom of dyspepsia | at 3 months, and 6 months
  Improvement of NDI-K, HADS,SEQ-FD at 3 and 6 months
Eradication of helicobacter pylori | at 3 months
  Eradication rate of helicobacter pylori at 3 months
Histologic finding of UGI tract | at initial and 3 months
  Change of accumulationof inflammatory cells, eosinophils of esophagus, stomachm duodenal mucosal biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Kee Wook Jung, MD, PhD, Principal Investigator — Asan Medical Center